CLINICAL TRIAL: NCT02237794
Title: Effect of Medical Treatment on Longitudinal Function of the Heart
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0049-14-HYMC
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Heart Function

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients Without Acute Heart Conditions: Patients without acute heart conditions who were hospitalized for other medical indications.

SUMMARY:
The purpose of this study is to determine the effect of medical treatment on longitudinal myocardial function. Patients who have been hospitalized for reasons other than heart disease will be examined with Transthoracic Cardiography before and after medical treatment to determine change in myocardial function.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients receiving above-mentioned medications

Exclusion Criteria:

* Patients suffering from heart conditions
* Patients unable to undergo Echocardiography
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in an Internal Medicine Department of the Hillel Yaffe Medical Center having a variety of medical conditions and treated with a variety of medications including Beta Blockers, Calcium Channel Blockers, Angiotensine Converting Enzyme Inhibitors and diuretics and do not suffer from overt heart conditions.
  --------------------------------------------------------------------------------
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Longitudinal Myocardial Function | Two Years
  Analysis of longitudinal contractility of the heart by the calculation of the heart's strain factor before and after chronic medication treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David Blondheim, MD, Study Chair — Hillel Yaffe Medical Center; Said Younis, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel